

# The effect of an opioid-free anesthetic on post-operative opioid consumption after laparoscopic bariatric surgery: a prospective, single-blinded, randomized controlled trial.

### CONSENT TO PARTICIPATE IN A RESEARCH STUDY

IRB Number: IRB19-051

**PRINCIPAL INVESTIGATOR:** Christine L. Oryhan, MD

Staff Anesthesiologist and Pain Physician

Virginia Mason Medical Center

1100 Ninth Avenue, MS: B2-AN Seattle WA 98101

**SUB-INVESTIGATOR (S):** Joseph Strunk, MD

Josiah Perez, MD Mohan Mallipeddi, MD

Lily Chang, MD Nam Nguyen, DO Shanley Deal, MD Angela Hirsh, MD

SUPPORTED BY: Department of Anesthesiology and Surgery

Virginia Mason Medical Center

**EMERGENCY CONTACT:** 911 – Medical Emergency

206-223-6980 (Day); 206-625-7373 (Night) Request to page Dr. Oryhan or Dr. Strunk

This is a clinical trial, a type of research study. Your study doctor will explain the clinical trial to you. Clinical trials include only people who choose to take part. Please take your time to make your decision about taking part.

This particular research in humans is designed by researchers at Virginia Mason Medical Center and is regulated by the Office of Human Research Protections (OHRP) and Food and Drug Administration (FDA).

Please note the following summary regarding your study participation. A more thorough explanation is available later in this document:



#### **STUDY SUMMARY**

You are being asked to take part in this study because you are going to receive a general anesthetic for your laparoscopic bariatric surgery. General anesthesia is used to put a person in a deep sleep so they don't feel pain during surgery.

The purpose of this study is to compare the postoperative pain control and postoperative opioid requirements of patients who, during bariatric surgery, received general anesthetic with no opioids to patients who received general anesthetic with opioids.

Your bariatric surgery will be performed as part of your standard care whether you are in the study or not. If you choose not to participate in the study, you and your doctor will discuss whether your anesthetic will or will not include opioids. If you do participate in the study, you will be randomly assigned (like flipping a coin) into one of two groups, but you won't be told which group you are in:

- Group A will receive anesthesia that includes Fentanyl, a type of opioid, for their bariatric surgery
- Group B will receive anesthesia with Dexmedetomidine, Ketamine, and esmolol, all drugs without opioids, for their bariatric surgery.

Fentanyl, Ketamine, and esmolol are approved by the U.S. Food and Drug Administration for use as part of a general anesthetic for the type of surgery you are receiving.

Dexmedetomidine is currently approved for certain anesthetic purposes, but its use in this study is investigational because the FDA has not approved its use as a general anesthetic for the type of surgery you are receiving. However, the safety profile of this drug as part of a general anesthetic has been well established in clinical trials.

If you participate in this study, researchers will:

- Evaluate your medical history to make sure you are eligible to participate
- Randomly assign you to either the group receiving anesthesia with opioids or to the group receiving anesthesia without opioids
- Collect information about your health before, during and after your bariatric surgery.
- Collect information about your pain and the pain medications you are prescribed as part of your normal care after your surgery.

Your participation is expected to last for about 3 months after your surgery so researchers can continue to access your medical records to follow how you are doing and what medications you are taking.

#### Risks:

- All general anesthetics have some risk of reaction to medications given.
- Opioids have risks that include slow breathing, constipation, slow return of intestinal function, confusion and sleepiness.
- Non-opioid anesthetics that may be used can also cause sleepiness, slow heart rate, and confusion.

#### Side effects:

 Pain after surgery varies between people. You may require supplemental IV or oral pain medications if your pain is not adequately managed.

There is a risk of loss of confidentiality of your information. You will read about the steps we take to help keep your information private and secure later in this form.

You are not expected to benefit personally from participating in this study, but we hope the information learned in this study will benefit other people in the future.

Taking part in this study is voluntary, and you may choose not to take part or may leave the study at any time. Choosing not to take part or leaving the study will not result in any penalty or loss of benefits to which you are entitled outside of this research.

# WHY IS THIS STUDY BEING DONE?

The purpose of this study is to evaluate whether a certain type of general anesthetic that avoids the use of opioids and uses other non-opioid medications provides similar postoperative pain control and postoperative opioid requirements as a more traditional general anesthetic that uses a limited amount of opioids.

This research is being done because we want to find the best way to provide pain relief and reduce the amount of opioids our patients need after bariatric surgery. Here at Virginia Mason Medical Center we have been providing a normal general anesthetic that uses a limited amount of opioids for this surgery for many years, but we want to know if we can offer the same pain relief by using non-opioid medications as a part of your general anesthesia. If we show that the two techniques are the same, then we can potentially make good pain control safer for all our patients having bariatric surgery.

### HOW MANY PEOPLE WILL TAKE PART IN THE STUDY?

About 196 people will take part in the study at Virginia Mason Medical Center.

# WHAT IS INVOLVED IN THE STUDY?

You will be "randomized" into one of two study groups described below. Randomization means you are put into a group by chance. It is like flipping a coin. A computer determines which group you are placed. Neither you nor the researcher will choose what group you will be in. You will not be told which group you are in. You will have an equal chance of being placed in any group.

- If you are in <u>Group A</u>: After we start your general anesthesia, you will receive a standard general anesthetic that includes a limited amount of Fentanyl, a type of opioid. Fentanyl is approved by the U.S. Food and Drug Administration for use as part of a general anesthetic for the type of surgery you are receiving.
- If you are in <u>Group B</u>: After we start your general anesthesia, you will receive no opioids until the recovery room. Your general anesthesia will include 3 non-opioid drugs, Dexmedetomidine, Ketamine, and esmolol. Ketamine and esmolol are all approved by the FDA for use as general anesthetic for the type of surgery you are receiving. Dexmedetomidine is currently approved for certain anesthetic purposes, but its use in this study is investigational because the FDA has not approved its use as a general anesthetic for the type of surgery you are receiving. However its safety profile as part of a general anesthetic has been well established in clinical studies.

# Before you begin the study ...

You will need to have the following exams, tests or procedures to find out if you can be in the study. These exams, tests or procedures may be done as part of your normal care even if you do not join the study. If you have had some of them recently, they may not need to be repeated. This will be up to your study doctor.

An evaluation of your medical history.

#### During the study ...

Your anesthesiologist caring for you in the operating room will determine the safest way to care for you during your surgery. They will explain this process and discuss all other anesthetic options with you prior to going to the operating room. After you fall asleep from general anesthesia, we will either use or avoid using opioids during your procedure. The other medications you receive as part of your anesthetic regimen will be the same, no matter which group you are in. It is important to note that your recovery room and subsequent care will not be different from the other study group—regardless of which arm you are randomized to, any pain you have after surgery will be treated the same.

The information generated from monitoring your health and the medications you take before, during and after the surgery will be used by the research team to help answer their study questions.

You will need these tests and procedures that are either being tested in this study or being done to see how the study is affecting your body.

Daily evaluation and examination while you remain inside the hospital

• Follow-up with your surgery team, as is described in the bariatric surgery pathway

If your surgeon decides during your surgery that it is necessary to perform the surgery as an open, and not laparoscopic procedure, you may stay in the study, however, you will no longer be assigned to a study group.

# **HOW LONG WILL I BE IN THE STUDY?**

You will be in the study for 3 months following surgery. You can stop participating in the study at any time. If you decide to stop being in the study, please talk to the researcher and your regular doctor first.

It is also possible your participation in the study will be ended by the research team, even if you want to remain in the study. This could happen, for example, if it is determined that participation is not in your best interest, or if the study is ended earlier than planned.

# WHAT ARE THE RISKS OF THE STUDY?

While on the study, we do not believe you will be exposed to any additional risks beyond what is already part of your standard of care. All general anesthetics have some risk of reaction to medications given. However, there may be risks we cannot predict. You should discuss this concern with the researcher and/or your regular doctor. Other procedures may be performed to make side effects less serious and uncomfortable. Many side effects go away shortly after the intervention is stopped, but in some cases side effects can be serious or long lasting or permanent.

Risks and side effects specific to the study group you are randomized to include:

Group A—Opioids have risks that include; slow breathing, constipation, slow return of intestinal function, confusion and sleepiness.

OR

➤ <u>Group B</u>—Non-opioid anesthetics that may be used can also cause; sleepiness, slow heart rate, and confusion.

#### Side effects:

➤ Pain after surgery varies between people. You may require supplemental IV or oral pain medications if your pain is not adequately managed. This will occur regardless of what group you are assigned.

There is also a risk of loss of confidentiality of your information. You will read about the steps we take to help keep your information private and secure later in this form.

For more information about risks and side effects, ask the researcher or contact Christine Oryhan, MD at 206-223-6980.

# **ARE THERE BENEFITS TO TAKING PART IN THE STUDY?**

If you agree to take part in this study, there will be no direct benefit to you. We hope the information learned from this study will benefit other people having bariatric surgery in the future.

# **WHAT OTHER OPTIONS ARE THERE?**

You may choose not to participate in this study. Instead of being in this study, you may choose to have the standard general anesthesia at the discretion of the anesthesiologist. Depending on your anesthesiologist's preference, you could receive an opioid restrictive general anesthetic, or an opioid free general anesthetic. The majority of general anesthetics for your type of surgery are currently carried out with limited opioid.

# WHAT ARE THE COSTS?

The costs of your bariatric surgery, including costs associated with general anesthetic, will be billed to your insurance, just as it would be if you were not in this study. Taking part in this study is not expected to lead to added costs to you or your insurance company. Please ask about any concerns regarding costs or insurance problems.

You will receive no payment for taking part in this study.

# WHAT IF YOU GET INJURED BECAUSE YOU TOOK PART IN THIS STUDY?

It is important you tell your study doctor, Christine Oryhan, MD if you feel you have been injured because of taking part in this study. You can speak with the doctor in person or call her at 206-223-6980.

You will get medical treatment if you are injured as a result of taking part in this study. Medical services will be offered at the usual charge and billed to your insurance. No funds have been set aside to compensate you in the event of injury. This does not limit your legal rights or ability to seek compensation for study related injuries.

#### WHAT ARE MY RIGHTS AS A PARTICIPANT?

Taking part in this study is voluntary, and you may choose not to take part or may leave the study at any time. Choosing not to take part or leaving the study will not result in any penalty or loss of benefits to which you are entitled outside of this research.

We will tell you about new information that may affect your health, welfare, or willingness to stay in this study.

# WHOM DO I CALL IF I HAVE QUESTIONS OR PROBLEMS?

 For questions about study procedures, study costs, or to report a study-related injury, contact the researcher Christine Oryhan, MD at 206-223-6980.  For questions about your rights as a research participant, contact the BRI Institutional Review Board (IRB) Manager at (206) 342-6916. The IRB Administrator manages the IRB, which is a group of people who review this research to protect your rights and welfare.

# Will I be notified if my data result in an unexpected or clinically relevant finding?

When data are collected and analyzed, there is the chance of finding something important or unexpected. There may be benefits to learning such results (such as early detection and treatment of a medical condition), but there are risks as well (such as feeling worried about a finding for which no treatment is required or appropriate).

In this study, you will be informed of any important or unexpected findings of possible clinical significance that may be discovered during review of results from your data. The results of your data will not be placed in your medical record with your primary care physician or otherwise.

The results from the data we collect in this research study are the same quality as what you would receive as part of your health care. As physicians who normally read the data we are collecting in this research, we will inform you if there are any important or unexpected findings so that you may discuss it with your primary care physician, although we do not expect this to be the case. However, if you believe you are having symptoms that may require care prior to receiving any information from this study, you should contact your primary care physician.

There are no plans to provide all participants with clinically relevant information from the research as a whole.

# STORAGE OF YOUR INFORMATION FOR POTENTIAL FUTURE RESEARCH:

We may store your information to use in future research. For future research with your information, researchers might remove identifiers, and the de-identified information might be used or shared with other researchers for future research without any additional consent from you. Findings or results from any testing or future research would not be reported back to you.

# WHERE CAN I GET MORE INFORMATION?

You will get a copy of this consent form and may also request a copy of the protocol (full study plan).

A description of this clinical trial will be available on *http://www.ClinicalTrials.gov*, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# AUTHORIZATION TO USE AND/OR DISCLOSE PROTECTED HEALTH INFORMATION FOR RESEARCH

We are required by special federal and state privacy laws to protect the privacy of your health information under the Health Insurance Portability and Accountability Act of 1996 (HIPAA) Privacy Rule. Researchers (investigators) would like to use your health information for research. This section describes what researchers will do with information about you. To learn more about your individual privacy rights, you may ask your provider for a Notice of Privacy Practices.

By signing this form, you authorize the individuals and entities listed below to use and disclose your health information for the purposes of the research study described in this form and in the above Consent ("Consent"). If you do not sign this form, then you will not be able to participate in this research study.

# WHAT IS PROTECTED HEALTH INFORMATION (PHI)?

PHI is information gathered by a health care provider, health plan, or researcher that identifies you or which includes facts that may tie your identity to your health record. PHI includes:

- Information from your existing or future medical records needed for this study as described in this form; and/or
- Information about you created during this study, as described above.
- This health information generally includes: demographics information, result of physical exams, histories and physicals, X-rays, diaries, questionnaires, records of treatments and side effects of treatments.

# WHO MAY USE OR SHARE MY PHI?

Virginia Mason and its health care providers, including but not limited to its primary care providers, are permitted to disclose your PHI to the Principal Investigator and Sub-Investigators (collectively, "Researchers") listed in the Consent. The Researchers may also use and disclose your health information between each other and with the other individuals and entities listed in this Authorization. In addition, the following health care providers may share your health information with the researchers.

- Virginia Mason Anesthesiologists.
- Virginia Mason Bariatric Surgeons.

#### WHAT MAY THE RESEARCHERS DO WITH MY PHI?

The researchers will use your health information to conduct the research. As part of the research they may share your information with certain people and groups. These may include:

- The sponsor of this study, the Department of Anesthesiology and Surgery at Virginia
  Mason Medical Center. The sponsor reviews the study and researchers must share some
  information with the sponsor.
- The Institutional Review Board (IRB) that approved this research, Benaroya Research Institute (BRI) IRB. The IRB reviews, audits, and monitors studies to protect the rights and safety of research participants.
- BRI Regulatory Compliance and Education Department in order to allow the Department to conduct routine internal quality reviews audits and monitor visits of the study and patient records.
- BRI coordinators, managers and assistants for the purposes of research study administrative and related support, including but not limited to pre-screening and follow up for research participants, and reporting to sponsors and government agencies.
- Federal and state agencies and their representatives that have oversight of the research study or to whom access is required under the law, which could include but are not limited to:
  - Food and Drug Administration (FDA)
  - Office for Human Research Protections (OHRP)
  - National Institutes of Health (NIH)
- Your health insurer(s) if they are paying for care provided as part of the research.

# **HOW WILL MY HEALTH INFORMATION BE KEPT PRIVATE?**

All efforts will be made to keep your personal information confidential; however, we cannot guarantee absolute confidentiality. Your personal information may be disclosed if required by law.

Researchers generally remove your name (and other information that could identify you) from your health information before sharing it. Once your PHI is given to a third party, that party may share it with someone else and the federal privacy law may no longer protect it; however, other privacy protections may still apply.

If research findings are published from this study, they will not identify you unless you allow it in writing.

### WHAT HAPPENS IF I WANT TO WITHDRAW MY AUTHORIZATION?

You may change your mind at any time and withdraw this authorization. This request must be made in writing to the investigator Christine Oryhan, MD at the address listed on page 1 of this form. Beginning on the date you withdraw, no new identifiable health information will be used for research. However, the researchers may continue to use and share the information that was provided before you withdrew your permission. If you withdraw your authorization, you will not be allowed to continue in this research study.

# **HOW LONG WILL THIS AUTHORIZATION LAST?**

This Authorization will expire 50 years from the date you sign it, unless you change your mind and revoke it in writing before then. The 50 year expiration date is because the information used and created during the study may be analyzed for many years, and it is not possible to know when this will be completed.

# PARTICIPANT'S CONSENT AND AUTHORIZATION

I have read and been given a chance to ask questions about this consent form and HIPAA authorization and agree to take part in this study. I will receive a signed copy of this consent form and HIPAA authorization.

| PARTICIPANT'S SIGNATURE | PAR | TICIPANT'S NA | AME (print) | DATE |
|---|---|---|---|---|
| CERTIFICATE OF PERSON OBTAINING I have provided an explanation of the above ask questions and request additional inform copy of this consent form has been given to | e research<br>nation rega | study, and have rding the study | | |
| SIGNATURE OF PERSON OBTAINING C | ONSENT | NAME OF PE | | AINING |
| DATE | | | | |
| WITNESS STATEMENT (complete only | if applicat | ole) | | |
| As an impartial third party, I witnessed the signature on this form. I attest that this en This person had enough time to consider t and voluntarily agreed to be in this study. | tire form w | as read to the p | oarticipant na | amed above. |
| Name of Witness (Print) | | | | |
| Signature of Witness | | | Date | |